CLINICAL TRIAL: NCT06330584
Title: Administration of Intranasal Midazolam for Anxiety in Palliative Care - a Double-blind, Randomized, Placebo-controlled Multicenter Exploratory Pilot Study With a Nested Pharmacokinetic Analysis
Brief Title: Administration of Intranasal Midazolam for Anxiety in Palliative Care
Acronym: AIM Care
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-00873
Record Dates: First submitted 2024-03-06; First posted 2024-03-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Acute Anxiety; Palliative Care
Keywords: Anxiety; Acute anxiety; Palliative Care; Midazolam; Nasal Spray
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled parallel-group multicenter exploratory pilot study with three study arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel except the personnel at the facility preparing the investigational medicinal product (IMP) (Hospital Pharmacy, University Hospital Basel), and all patients will be blinded to the assigned treatment. Allocation will be concealed using sequentially coded drug packs (using consecutive patient identification numbers from 1 to 36) containing the IMP that are otherwise identical. Each drug pack will contain two nasal sprays of identical appearance. Patients and all trial personnel involved in recruitment and care of patients, trial assessment, monitoring, and analyses will be blinded to the assigned trial arm. Blinding will be upheld until the last patient (36 patients, i.e., 12 per study arm) has completed the pilot study and data entry into the trial database has been completed.
  To safeguard blinding, placebo formulation will be produced with the same pH as the active study drug formulations to mimic nasal irritation induced by verum sprays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Total dose of midazolam = 0 mg (no active compound)
  Interventions: Drug: Placebo Nasal Spray 0 mg/spray
- Standard of Care (SOC) (Active Comparator): Total dose of midazolam = 0.9 mg
  Interventions: Drug: Midazolam Nasal Spray 0.45 mg/spray
- Double Dose of Standard of Care (2xSOC) (Active Comparator): Total dose of midazolam = 1.8 mg
  Interventions: Drug: Midazolam Nasal Spray 0.9 mg/spray

INTERVENTIONS:
Drug: Placebo Nasal Spray 0 mg/spray — A unit-dose nasal spray will be used for the intervention.
  1 spray (= 0.1 μl = 0 mg midazolam/spray) in each nostril, i.e., no active compound
  Arms: Placebo
Drug: Midazolam Nasal Spray 0.45 mg/spray — A unit-dose nasal spray will be used for the intervention.
  1 spray (= 0.1 μl = 0.45 mg midazolam/spray) in each nostril, i.e., total dose of midazolam 0.9 mg
  Arms: Standard of Care (SOC)
Drug: Midazolam Nasal Spray 0.9 mg/spray — A unit-dose nasal spray will be used for the intervention.
  1 spray (= 0.1 μl = 0.9 mg midazolam/spray) in each nostril, i.e., total dose of midazolam 1.8 mg
  Arms: Double Dose of Standard of Care (2xSOC)

SUMMARY:
The goal of this double-blind, randomized, placebo-controlled parallel-group multicenter exploratory pilot study (three study arms) is to describe effects and safety of different doses of intranasal midazolam to treat acute anxiety in palliative care patients, while providing pharmacokinetic and pharmacodynamic data.

DETAILED DESCRIPTION:
36 patients (12 per study arm) will be enrolled. All patients hospitalized at the four study sites, which are prescribed intranasal midazolam in their as-needed drug regimen and who meet inclusion criteria, are eligible. Patients will be asked for consent at the time of prescription of midazolam by the attending physician. Patients who have provided consent and have been randomized to one of the arms will be included (block randomization).

In a nested analysis, pharmacokinetic properties of all three doses will be analyzed in participants with available venous access.

The primary outcome is the change in patient-reported levels of anxiety from baseline. Secondary outcomes include time until first requested additional dose, cumulative number of doses including time points of administration after the first application, oxygen saturation, heart rate, cortisol levels in oral fluid, levels of sedation on the Richmond Agitation Sedation Scale Palliative Version (RASS-PAL), and occurrence of (serious) adverse events.

The primary and secondary outcomes will be assessed at baseline, i.e., immediately before the intervention (0 minutes) and 30 minutes after the intervention. The secondary outcomes 'Time to first requested additional dose' and 'Cumulative number of doses over 24 hours' as well as (serious) adverse events will be assessed starting 30 minutes after the intervention up to 24 hours after the intervention.

In patients included in the nested pharmacokinetic analysis, basic pharmacokinetic parameters will additionally be assessed at 10 time points, starting at baseline (0 minutes) up to 240 minutes after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult palliative care patients (≥ 18 years) hospitalized at one of the study sites
* Self-reported acute anxiety with clinical indication for intranasal midazolam administration according to attending physician
* Patient willing and able to provide written informed consent
* Informed consent as documented by signature
* Patient willing and able to complete anxiety assessment
* Additionally for nested pharmacokinetic analysis: Patients with available central or peripheral venous access, i.e., peripheral venous catheter (PVC), central venous catheter (CVC), peripherally inserted central venous catheter (PICC) line, midline catheter, or PORT-A-CATH® (PAC), and patient willing and able to provide blood samples

Exclusion Criteria:

* Intranasal midazolam prescribed for seizures
* Midazolam (any route of administration) prescribed and administered for continuous sedation
* History of allergy or hypersensitivity to midazolam
* History of benzodiazepine-related paradoxical reaction to midazolam
* Acute narrow-angle glaucoma
* Impaired nasal absorption (e.g., nasogastric tube, nasal obstruction, nasal polyps, etc.)
* Intranasal midazolam within 24 h before study enrollment
* Time between informed general consent for study participation through investigators and planned midazolam administration < 24 h
* Co-medication with strong CYP3A4 inducers or inhibitors according to pre-defined list (FDA)
* Recently initiated therapy with strong opioids (i.e., within past 5 days)
* Co-medication with other CNS depressants causing clinically relevant degree of sedation
* Inability to follow the procedures of the study (i.e., provision of Informed Consent, completion of assessment tool, e.g., due to language problems or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in anxiety levels, measured by Visual Analogue Scale (VAS) and quantified by Numerical Rating Scale (NRS) | t [0 minutes, 30 minutes]
  Patient-reported levels of anxiety, measured by VAS (0-100 mm, from left 'no anxiety at all' to right 'worst possible anxiety') at baseline (0 minutes) and 30 minutes after study drug or placebo administration. The VAS response will be quantified measuring the distance in mm from zero to the position of the VAS response on a ruler (=100 mm, separated by 1 mm intervals), with 0 mm representing absence of anxiety, and 100 mm representing maximal possible anxiety.

SECONDARY OUTCOMES:
Sedation | t [0 minutes, 30 minutes]
  Richmond Agitation Sedation Scale Palliative Version (RASS-PAL)
  The RASS-PAL ranges from +4 (combative) to -5 (not rousable), where a higher score (below 0) is associated with agitation and a lower score (below 0) is associated with sedation. A score of 0 (alert and calm) is considered the most balanced state.
Oxygen saturation SaO2 (percent %) | t [0 minutes, 30 minutes]
  Oxygen saturation
Heart rate (bpm) | t [0 minutes, 30 minutes]
Cortisol levels in oral fluid | t [0 minutes, 30 minutes]
Time to first requested additional dose | t [starting assessment 30 minutes after intervention up to 24 hours after intervention]
  30 minutes after the intervention, additional doses may be administered as-needed. The time point until the first additional dose starting 30 minutes after the intervention is assessed. The time point can occur anywhere between 30 minutes and 24 hours after the intervention.
Cumulative number of doses over 24 hours | t [starting assessment 30 minutes after intervention up to 24 hours after intervention]
  As additional doses may be administered after 30 minutes after the intervention, every additional requested dose is assessed and the total number of doses over 24 hours after the intervention is calculated.
Number of patients with adverse drug events (ADEs) | t [starting immediately after intervention up to 24 hours after intervention]
  The adverse drug reactions (ADRs, i.e. reactions to be expected from the intervention based on clinical experience and the SmPC of Nayzilam), and (serious) adverse events ((S)AEs) will be assessed at three different time windows: between study drug administration and 30 minutes after the intervention, 30 minutes after study drug administration, and up to 24 hours after the intervention.
Peak plasma concentration (Cmax) | t [0 minutes up to 240 minutes after intervention]
  Pharmacokinetic parameter obtained by non-compartmental analysis (NCA) or compartmental analysis (CA) in a pre-defined eligible subset of patients (i.e., patients with a central or peripheral venous access).
  There will be 10 measurement points: at baseline (0 minutes, i.e., before intervention) and at t [2.5, 5, 10, 15, 30, 60, 120, 180, 240 minutes].
Time to reach the peak plasma concentration (Tmax) | t [0 minutes up to 240 minutes after intervention]
  Pharmacokinetic parameter obtained by non-compartmental analysis (NCA) or compartmental analysis (CA) in a pre-defined eligible subset of patients (i.e., patients with a central or peripheral venous access).
  There will be 10 measurement points: at baseline (0 minutes, i.e., before intervention) and at t [2.5, 5, 10, 15, 30, 60, 120, 180, 240 minutes].
Elimination half-life (t1/2) | t [0 minutes up to 240 minutes after intervention]
  Pharmacokinetic parameter obtained by non-compartmental analysis (NCA) or compartmental analysis (CA) in a pre-defined eligible subset of patients (i.e., patients with a central or peripheral venous access).
  There will be 10 measurement points: at baseline (0 minutes, i.e., before intervention) and at t [2.5, 5, 10, 15, 30, 60, 120, 180, 240 minutes].
Area under the curve (AUC0-Τ, AUC0-∞) | t [0 minutes up to 240 minutes after intervention]
  Pharmacokinetic parameter obtained by non-compartmental analysis (NCA) or compartmental analysis (CA) in a pre-defined eligible subset of patients (i.e., patients with a central or peripheral venous access).
  There will be 10 measurement points: at baseline (0 minutes, i.e., before intervention) and at t [2.5, 5, 10, 15, 30, 60, 120, 180, 240 minutes].

CONTACTS AND LOCATIONS:
Overall Officials: Carla Meyer-Massetti, PhD, Study Chair — Inselspital, Universitätsspital Bern
Locations (5):
- Switzerland (5):
  - Palliativzentrum Bethesda Spital, Basel, Canton of Basel-City
  - Inselspital, Universitätsspital Bern, Bern
  - Universitäres Zentrum für Palliative Care (UZP), Bern
  - Zentrum für Palliative Care, Stadtspital Zürich, Zurich
  - Kompetenzzentrum Palliative Care, Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No